CLINICAL TRIAL: NCT02355509
Title: Effect of Acarbose on Postprandial Lipoprotein Levels in Glucose Intolerant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Francisco J. Gómez Pérez, Chief of the Department of Endocrinology and Metabolism, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REF.1467
Record Dates: First submitted 2015-01-21; First posted 2015-02-04 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Glucose Intolerance; Postprandial Hyperglycemia; Cardiovascular Risk Factor
Keywords: Acarbose; Postprandial lipemia; Cardiovascular risk
MeSH Terms: conditions — Glucose Intolerance; Hyperglycemia | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A placebo drug is given for three months
  Interventions: Drug: Placebo
- Acarbose (Experimental): Acarbose is given for three months
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Acarbose — Acarbose dose was progressively titrated (50 mg/day per week up to 150 mg/day) to reduce the known adverse effects of acarbose such as flatulence, bloating, diarrhea, abdominal pain.
  The treatment for three months
  Other Names: Glucobay
  Arms: Acarbose
Drug: Placebo — Placebo pills are given instead of acarbose in this group
  Arms: Placebo

SUMMARY:
Is a randomized, double-blind, placebo-controlled trial to determine the behavior of hyperglycemia and postprandial lipemia after a standard mixed meal load in patients with carbohydrate intolerance treated with acarbose.

DETAILED DESCRIPTION:
To gather our patients, we invite the relatives of diabetic patients seen at the endocrinology consultation to participate in the study.

* Patients are placed into an isocaloric diet for 4 weeks before the study and are advised not to change their baseline physical activity.
* Patients are randomized to receive acarbose or placebo for 3 months blinded to investigators and patients.
* Acarbose dose is progressively titrated (50 mg/day per week up to 150 mg/day) to reduce the known adverse effects of acarbose such as flatulence, bloating, diarrhea, abdominal pain.
* In each subject, a 5-hr-postprandial mixed meal test is performed at baseline and after assigned treatment was completed. Glucose, insulin, triglycerides and total cholesterol were measured at 0, 5, 10, 20, 30, 60, 120, 180, 240 and 300 minutes after the mixed meal load. Apo B was measured by nephelometry and oxLDL using a monoclonal antibody 4E6 based competition (ELISA assay, Mercodia) at 0 and 300 minutes.
* The standard mixed meal load, a 470 kcal breakfast, (47.76% carbohydrate, 22.66% proteins, 29.58% fat), consisted of: 1 sandwich (prepared with 50 g of Savory´s™ turkey breast ham, 30 g of Savory´s™ panela cheese, 2 tablespoons of Hellmann's™ mayonnaise and 2 slices of Bimbo´s™ white bread), 100 g of Red DeliciousTM apple and 250 mL of Alpura´s™ lactose-free, light milk.
* During the 3-month treatment, patients have 3 follow-up monthly consultations to evaluate weight gain and treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of carbohydrate intolerance according to the WHO criteria, without any treatment.

Exclusion Criteria:

* patients with BMI >32 kg/m2, triglycerides and/or total cholesterol > 300 mg/dl, known renal, liver or gastrointestinal disease and positive smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in postprandial oxLDL | 3 months treatment
  In each subject oxLDL is measured using a monoclonal antibody 4E6 based competition (ELISA assay, Mercodia) at 0 and 300 minutes in a postprandial 5 hour test, pre and post-treatment

SECONDARY OUTCOMES:
Chance in postprandial hyperglycemia | 3 months treatment
  A 5 hour postprandial test is performed in each patient, were glucose is measured at 0, 5, 10, 20, 30, 60, 120, 180, 240 and 300 minutes, pre and post-treatment
Chance in postprandial insulin levels | 3 months treatment
  A 5 hour postprandial test is performed in each patient, were insulin is measured at 0, 5, 10, 20, 30, 60, 120, 180, 240 and 300 minutes, pre and post-treatment
Change in LDL concentration | 3 months treatment
  We measure basal LDL concentration in each patient, pre and post-treatment
Change in HDL concentration | 3 months treatment
  We measure basal HDL concentration in each patient, pre and post-treatment
Change in Apolipoprotein B (ApoB) concentration | 3 months treatment
  In each subject ApoB is measured, using nephelometry, at 0 and 300 minutes in a postprandial 5 hour test, pre and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fracisco J Gómez-Pérez, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición, Salvador Zubirán, Mexico City, Mexico City, Mexico